CLINICAL TRIAL: NCT07068139
Title: The Role of Artificial Intelligence in Predicting Stage and Survival in Non-Small Cell Lung Cancer
Brief Title: AI-Based Prediction of Stage and Survival in Non-Small Cell Lung Cancer: A Retrospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Hilkat Fatih Elverdi (Other)
Responsible Party: Sponsor-Investigator, Hilkat Fatih Elverdi, Thoracic Surgery Resident, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/194-318
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer; Artificial Intelligence (AI) in Diagnosis
Keywords: Non-Small Cell Lung Cancer; Artificial Intelligence; Deep Learning; Radiology; Thoracic Surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC Surgery Cohort: This cohort includes patients who were diagnosed with non-small cell lung cancer (NSCLC) and underwent surgical treatment at Ondokuz Mayis University Hospital. Preoperative PET-CT and chest CT images and corresponding postoperative histopathological data were retrospectively collected and analyzed to develop an artificial intelligence model for predicting tumor stage and survival.
  Interventions: Other: AI-Based Predictive Modeling

INTERVENTIONS:
Other: AI-Based Predictive Modeling — This is not a therapeutic or diagnostic intervention. The study uses a retrospective dataset of radiologic and pathological records to train and validate a deep learning model designed to predict tumor stage and survival in patients with non-small cell lung cancer (NSCLC). No experimental procedure is applied to participants.
  Other Names: Deep Learning Algorithm, Retrospective Imaging Analysis

SUMMARY:
This study aims to evaluate the role of artificial intelligence (AI) in predicting disease stage and survival in patients diagnosed with non-small cell lung cancer (NSCLC). Using a retrospective design, the research will analyze radiologic imaging data (PET-CT and chest CT) and corresponding histopathological results of patients who underwent lung cancer surgery at Ondokuz Mayis University Hospital.

The goal is to develop and validate a deep learning-based AI model that can automatically assess preoperative radiologic features and estimate postoperative tumor stage and survival outcomes. By integrating radiologic data with confirmed pathological diagnoses, the AI system is expected to provide clinical decision support that can improve diagnostic speed, reduce human error, and help clinicians predict prognosis more accurately.

This study does not involve any experimental treatment or prospective follow-up of patients. All data will be collected from existing medical records. The findings may contribute to the digital transformation of healthcare and promote the use of AI tools in thoracic oncology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosed with non-small cell lung cancer (NSCLC)
* Underwent surgical treatment for NSCLC at Ondokuz Mayis University Hospital
* Available preoperative PET-CT and chest CT imaging
* Available postoperative histopathological diagnosis and staging
* Signed informed consent form for data use in research

Exclusion Criteria:

* Age < 18 years
* No available PET-CT or chest CT imaging in hospital records
* No available histopathological diagnosis in hospital records
* Diagnosed with a type of lung cancer other than NSCLC
* Patients who did not undergo surgery
* Patients who did not provide informed consent for retrospective data use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients who underwent surgical treatment for non-small cell lung cancer (NSCLC) at Ondokuz Mayis University Hospital in Samsun, Türkiye. Eligible patients are selected from the hospital's electronic medical records and radiologic imaging archive between January 2010 and March 2025. The population reflects a clinical sample from a tertiary referral center serving a diverse adult patient population in the Black Sea region of Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Development of AI Model for Predicting Tumor Stage and Survival | From data extraction to completion of model training and validation (estimated by September 2025)
  The primary outcome of this study is to develop and validate a deep learning-based artificial intelligence model that can predict postoperative tumor stage and survival in patients with non-small cell lung cancer using preoperative PET-CT and chest CT imaging data. The primary outcome will be considered achieved when at least 80% of the planned patient dataset (150 patients) has been successfully included and used for model development.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (e.g., imaging features, demographic variables, survival outcomes) may be shared for academic and research purposes upon reasonable request and following institutional data-sharing agreements. No personal identifiers will be included.